CLINICAL TRIAL: NCT05708820
Title: Online Education Programme for People With Type 1 Diabetes and Suboptimal Metabolic Control
Acronym: OPTIM@TE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Mutua de Terrassa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: EO2014
Record Dates: First submitted 2022-03-29; First posted 2023-02-01 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Diabetes Mellitus, Type I
Keywords: Diabetes Mellitus, Type I; education programme; online
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care (Active Comparator): Group in face-to-face session
  Interventions: Behavioral: Standard education programme
- Online education programme (Experimental): Group in online sessions
  Interventions: Behavioral: Online education programme

INTERVENTIONS:
Behavioral: Online education programme — Online group will follow the education programme through videos that they can view at any time and a live session to answer questions.
  Arms: Online education programme
Behavioral: Standard education programme — Face-to-face educacion programme in a group session
  Arms: Standard care

SUMMARY:
The aim of this study is to evaluate the effectiveness of an online intervention for people with type 1 diabetes who present not optimal control of the disease.

DETAILED DESCRIPTION:
Study area: adults with type 1 diabetes, HbA1c >7.5%, >3 years diagnosed. Methods: randomized clinical trial. It will include 60 participants . The improvement of Glycated Haemoglobin in both groups before and after intervention will be compared; adherence to the treatment, quality of life, time in the glycaemic range, perception of hypoglycaemia and knowledge about diabetes.

ELIGIBILITY:
Inclusion Criteria:

* HbA1c ≥7,5%
* More than 3 years of diagnosis
* Ability to follow online sessions
* Having a device to follow up the education programme

Exclusion Criteria:

* Pregnants
* People on corticosteroid treatment
* People with severe disease
* People with continuous subcutaneous insulin infusion (CSII)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-12-14 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
HbA1c | Change from Baseline at 12 months
  glycosylated hemoglobin

SECONDARY OUTCOMES:
Time in Range (TIR) | Change from Baseline at 12 months
  Time spent between 70-180 mg/dl measured by glucose sensor
Knowledge related to diabetes management | Change from Baseline at 12 months
  Diabetes Knowledge Questionnaire (DKQ2)- 15 questions with 4 options, high score indicates maximum level of knowledge
Awareness of hypoglycemia | Change from Baseline at 12 months
  Clarke Test- 8 questions, ≥ 4 answers with R= reduced awareness

CONTACTS AND LOCATIONS:
Overall Officials: Núria Alonso, RN, Principal Investigator — Hospital Universitari Mútua Terrassa
Locations (2):
- Spain (2):
  - Hospital Mutua de Terrassa, Terrassa, Barcelona
  - Hospital Universitari Mútua de Terrassa, Terrassa, Barcelona

IPD SHARING:
Plan to Share IPD: No